CLINICAL TRIAL: NCT01766934
Title: Non-interventional, Prospective, Long-term Safety Data Collection of Zarzio® / Filgrastim HEXAL® in Healthy Unrelated Stem Cell Donors Undergoing Peripheral Blood Progenitor Cell Mobilization
Brief Title: Non-interventional, Long-term Safety Data Collection of Zarzio® / Filgrastim HEXAL® in Stem Cell Donors
Acronym: SMART
Status: Completed | Type: Observational
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Other Study IDs: EP06-501
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hematopoietic Stem Cell Mobilization
Keywords: Peripheral blood progenitor cell mobilization; allogenic hematopoetic stem cell transplantation; recombinant human granulocyte colony stimulating factor; filgrastim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Data collection on the safety and efficacy of Zarzio® / Filgrastim HEXAL® in adult healthy unrelated stem cell donors undergoing peripheral blood progenitor cell mobilization.

DETAILED DESCRIPTION:
This will be a prospective, non-interventional long term data collection study. Adult healthy unrelated stem cell donors receiving Sandoz' filgrastim according to the stem cell mobilization protocols of the respective apheresis centers will be monitored for safety and efficacy during the mobilization period, and a systematic safety data follow-up will be implemented for up to 10 years after mobilization.

ELIGIBILITY:
Inclusion Criteria:

Volunteer adult healthy unrelated donors who have received at least one dose of Sandoz' filgrastim for PBPC mobilization

Exclusion Criteria:

* Donors of age <18 years
* Related to recipient
* Chronic significant organ diseases
* Systemic autoimmune diseases
* Chronic infectious diseases
* History of malignant disease
* Pregnant and breastfeeding women
* Hypersensitivity to E. coli derived proteins
* Hypersensitivity to the active substance or to any of the excipients of Sandoz' filgrastim
* Absolute and relative contraindications as specified in the SmPC of Sandoz' filgrastim
* Participation in previous stem cell mobilization procedures
* Previous or concurrent use of other mobilizing agents, e.g. plerixafor
* Informed consent was not signed prior to beginning of documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult, unrelated, healthy volunteers who received at least one dose of Sandoz' filgrastim
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2011-05; Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Incidence of drug-related adverse events following mobilization with Sandoz' filgrastim. | each patient will be followed for 10 years after mobilization
  The primary objective is to investigate adverse events that are suspected to be related to stem cell mobilization with the Sandoz' filgrastim in healthy unrelated donors.

SECONDARY OUTCOMES:
Efficacy assessment in terms of the CD34+ cell count. | CD34+ cells are counted on 1 day immediately preceding apheresis
  The secondary objective is to investigate the efficacy of stem cell mobilization with the Sandoz' filgrastim in terms of the CD34+ cell count.

CONTACTS AND LOCATIONS:
Overall Officials: Hexal AG, Study Chair — Hexal AG
Locations (2):
- Germany (2):
  - German Red Cross Blood Donor Service Baden-Wuerttemberg-Hessen, Institute for Transfusion medicine und Immunohematology Frankfurt am Main, Frankfurt am Main, Hesse
  - German Red Cross Blood Donor Service Baden-Wuerttemberg-Hessen, Institute for Clinical Transfusion medicine and Immunogenetics Ulm (IKT), Ulm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heyn J, Brauninger S, Dimova-Dobreva M, Mathieson N, Koptelova N, Kolpakova A, Seidl C, Reinhardt P, Tsamadou C, Schrezenmeier H, Nakov R, Seifried E, Bonig H. Superior physical and mental health of healthy volunteers before and five years after mobilized stem cell donation. J Transl Med. 2022 Mar 14;20(1):121. doi: 10.1186/s12967-022-03322-w. PMID 35287672